CLINICAL TRIAL: NCT05376384
Title: Ovarian Cyst's Enucleation Spillage Score. An Observational Study of Cyst Characteristics for Spillage During Laparoscopic Enucleation
Brief Title: Ovarian Cyst's Enucleation Spillage Score
Acronym: OC-ESS
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Carlo Ronsini, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 0013958/i-
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cysts; Spillage
Keywords: ovarian cysts; laparoscopy; cyst enucleation; spillage
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients, over 18 years old, undergoing laparoscopic cyst enucleation surgery with an occasional, unanticipated finding of cyst rupture and intraoperative spillage
  Interventions: Diagnostic Test: ultrasound parameters; Procedure: intraoperative parameters
- Control: Patients, over 18 years old, undergoing laparoscopic cystic enucleation surgery with the extraction of the intact operative specimen.
  Interventions: Diagnostic Test: ultrasound parameters; Procedure: intraoperative parameters

INTERVENTIONS:
Diagnostic Test: ultrasound parameters — Annotation of ultrasonographic features of ovarian cyst. The parts examined are size, laterality, content, margins, and color score.
Procedure: intraoperative parameters — Annotation of intraoperative features of ovarian cyst. The characteristics under review are: surgeon experience, previous surgery, adhesions, and uterine manipulator use

SUMMARY:
Cystic enucleation is one of the most common conservative surgeries in gynecology; it is commonly performed by a minimally invasive approach such as laparoscopy. A high percentage of these surgeries (6-88 % of cases) are complicated by the cystic rupture with intra-abdominal spillage of its contents (spillage). This occurrence affects the surgical and prognostic outcome by lengthening the time of surgery, increasing the risk of postoperative infection or granulomatous peritonitis, of possible second manifestation of the pathology (example: endometriosis), and in the case of neoformation of a carcinomatous nature by leading to an increase in the stage of disease, exposing patients to a prognostic disadvantage and the need for adjuvant treatments also avoidable. In addition, the previous spillage may be associated with the adherent syndrome with repercussions on patients' morbidity and fertility. For these reasons, it is crucial to optimize the selection of patients who are candidates for cystic enucleation.

The present study aims to evaluate a series of ultrasound, medical history, and surgical-preoperative parameters to develop a predictive score for the risk of spillage during laparoscopic surgery. Prospective Observational Study. The study aims to enroll 156 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Patients undergoing laparoscopic cystic enucleation
* Patients who underwent pelvic ultrasound examination within 30 days prior to surgery
* Patients who signed informed consent for the study
* ECOG performance status < 2

Exclusion Criteria:

* Pregnancy status
* Patients with cardiological, neurological, or metabolic disorders not treated pharmacologically
* ASA III
* Patients undergoing laparotomy conversion prior to enucleation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Naples Metropolitan area, southern Italy, where our university hospital is located, suffering from adnexal cystic neoformation for which they need to undergo laparoscopic cystic enucleation surgery. Patients will receive the standard of care regardless of participation in the study, in which they will participate voluntarily and after signing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Spillage Rate | 12 months
  Identification of spillage rate during laparoscopic cystic enucleation in patients with the risk factors considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi della Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No